CLINICAL TRIAL: NCT00778128
Title: A Phase I Clinical Study of Oral CP-4126 in Patients With Advanced Solid Tumour
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clavis Pharma (Industry)
Responsible Party: Trygve Bergeland, Clavis Pharma ASA
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP4126-111
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2010-09

CONDITIONS: Solid Tumors
Keywords: CP-4126; Cancer; Metastatic; Solid tumours; Gemzitabine; Gemzar
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — CP 4126; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Step 1: Dose escalation - oral CP-4126
  Step 2: Oral CP-4126 on day 1 and 15 in a 4 week schedule. One dose (only) gemcitabine IV on day 8.
  Interventions: Drug: CP-4126; Drug: Gemcitabine
- 2 (Experimental): Step 1: Dose escalation - oral CP-4126
  Step 2: Oral CP-4126 on day 8 and 15 in a 4 week schedule. One dose (only) gemcitabine IV on day 1.
  Interventions: Drug: CP-4126; Drug: Gemcitabine

INTERVENTIONS:
Drug: CP-4126 — Step 1: Dose escalation oral CP-4126 until maximum tolerated dose. Step 2: Oral CP-4126 day 1 and 15 + IV Gemcitabine 1000 mg/m2 day 8 in a 4 week schedule until complete response or disease worsening / progression
Drug: Gemcitabine — Step 1: Dose escalation oral CP-4126 until maximum tolerated dose Step 2: Oral CP-4126 day 8 and 15 + IV Gemcitabine 1000 mg/m2 day 1 in a 4 week schedule until complete response or disease worsening / progression

SUMMARY:
At step 1, patients with advanced solid tumors will receive CP-4126 capsules following a dose escalation schedule until the maximum tolerated dose is reached. At step 2, 20 patients will be randomized. They will receive at days 1 and 8 in a double cross design either oral CP-4126 at the recommended dose or gemcitabine 1000mg/m2 intravenously. At both steps, the schedule of treatment will be day 1, 8, 15 q4w until complete response or disease worsening/ progressing. All further treatment at step 2 will be oral CP-4126.

DETAILED DESCRIPTION:
This is a multicentre clinical study conducted in Belgium and in The Netherlands. The study is a phase I divided in 2 steps: The first step is a dose escalation to define the RD. At the second step the PK profile of oral CP-4126 will be compared with the PK profile of IV gemcitabine. In addition, the study is conducted to characterize the tolerability of oral CP-4126, to evaluate its bioavailability, and to make a preliminary assessment of antitumor activity in patients with solid tumours.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed solid tumour diagnosis
2. Locally advanced or metastatic disease, for which there is no known effective treatment
3. Performance Status 0 - 2 according to ECOG (Eastern Cooperative Oncology Group) Performance Status
4. Age 18 years or more
5. Life expectancy > 3 months
6. Adequate hematological and biological functions:
7. Signed informed consent

Exclusion Criteria:

1. Symptomatic brain metastases
2. Current peripheral neuropathy of grade > 1 according to the National Cancer Institute (NCI) - Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0
3. Radiotherapy

   * to more than 30 % of bone marrow
   * single dose up to 8 Gy
   * less than one week prior to the study treatment
   * of the upper GI tract
4. Mucositis of the upper digestive tract, including stomatitis
5. Participation in another therapeutic clinical study within 30 days of enrolment or during this clinical study
6. Previous anticancer therapy (chemotherapy, hormone therapy or immunotherapy) within 30 days prior to the first dose of oral CP-4126 [6 weeks for mitomycin C and BCNU (= carmustine) and CCNU (=lomustine)]
7. Requirement of concomitant treatment with a non-permitted medication including alternative drugs and high doses of vitamins
8. History of allergic reactions to gemcitabine
9. Presence of any serious concomitant systemic disorders incompatible with the clinical study (e.g. uncontrolled inter-current illness including ongoing or active infection)
10. Presence of any significant central nervous system or psychiatric disorder(s) that would hamper the patient's compliance
11. Pregnant or breast feeding women
12. Absence of adequate contraception for both male and female fertile patients for the duration of the study; and also for six months after last treatment
13. Known positive status for HIV and/or hepatitis B or C
14. Any reason why, in the investigator's opinion, the patient should not participate
15. Condition that impairs ability to swallow pills
16. Coeliac disease or any other lipid malabsorption syndrome
17. Drug and/or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Step 1: MTD of oral CP-4126 in patients with advanced solid tumours, followed by establishing the recommended dose | 6 months
Step 2: Pharmacokinetic parameters comparison of oral CP-4126 with IV gemcitabine | 12 months

SECONDARY OUTCOMES:
Tolerability of oral CP-4126 | 12 months
Biovailability of oral CP-4126 | 12 months
Preliminary assessment of antitumor activity of oral CP-4126 | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad H Awada, MD, Principal Investigator — Institute Jules Bordet
Locations (3):
- Institute Jules Bordet, Brussels, Belgium
- Netherlands (2):
  - The Netherlands Cancer Institute, Amsterdam
  - University Medical Centre Utrecht, Utrecht

REFERENCES:
- [Derived] Stuurman FE, Voest EE, Awada A, Witteveen PO, Bergeland T, Hals PA, Rasch W, Schellens JH, Hendlisz A. Phase I study of oral CP-4126, a gemcitabine derivative, in patients with advanced solid tumors. Invest New Drugs. 2013 Aug;31(4):959-66. doi: 10.1007/s10637-013-9925-z. Epub 2013 Jan 24. PMID 23345000